CLINICAL TRIAL: NCT07202065
Title: Role of Antibiotic Therapy or Immunoglobulin On iNfections in hAematoLogy (Dose-Ig)
Brief Title: Role of Antibiotic Therapy or Immunoglobulin On iNfections in hAematoLogy Dosing Immunoglobulin (Dose Ig)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRU-RPT-22 Dose-Ig
Record Dates: First submitted 2025-09-24; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Myeloma; Non Hodgkin's Lymphoma; Leukemia
Keywords: immunoglobulin; antibiotics; myeloma; leukaemia; lymphoma; non Hodgkins; infection; infections; blood; cancer; haematology
MeSH Terms: conditions — Neoplasms, Plasma Cell; Leukemia; Lymphoma; Infections; Neoplasms | interventions — gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Up to 900 participants will be recruited to the RATIONAL-PT, including up to 300 per domain. The aim of the platform is to determine optimal supportive care interventions for patients with haematological malignancies. The primary outcome for the platform is Event-free survival (EFS), defined as time from randomisation (or, in domains with a single treatment arm, time from registration) until occurrence of a Grade 3 or higher infection (as defined by CTCAE Version 5), or death from any cause. Data from each domain will contribute to the primary analysis.
Masking Description: An independent outcome adjudication committee will meet to review and adjudicate infection outcome data. These committee members will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Low dose (IgRT) immunoglobulin replacement therapy (Other): Participants will be treated with intravenous immunoglobulin monthly (every 4 weeks ± 1 week) at a dose of 0.25g/kg. No dose adjustment for trough serum (IgG) immunoglobulin G levels is required.
  Interventions: Biological: Immune Globulin Intravenous
- Arm B: Usual dose (Other): Participants will be treated with intravenous immunoglobulin monthly (every 4 weeks ± 1 week) at a dose of 0.4g/kg, modified to achieve an IgG trough level of at least lower limit of age-specific serum (IgG) immunoglobulin G reference range.
  Interventions: Biological: Immune Globulin Intravenous

INTERVENTIONS:
Biological: Immune Globulin Intravenous — Participants will be treated with intravenous immunoglobulin monthly (every 4 weeks ± 1 week).
  Other Names: IVIG

SUMMARY:
This study is being conducted to find out how safe and effective different strategies of infection prevention are in comparison to each other, for preventing infection in patients with blood cancers. The best way to find out this information is to directly compare the effect of different treatment strategies in patients with blood cancers. We want to know how these different treatments impact on your health and your use of healthcare services.

This research project uses an Adaptive Platform Design. This design allows the researchers to compare multiple infection prevention strategies within the same trial at the same time (rather than running separate trials), to analyse results as the trial occurs and to add new research questions during the course of the trial.

The treatments that you may receive as part of the study will be determined by which domain(s) of the platform you participate in. By combining data collected within each domain as part of the platform, the researchers can investigate and compare treatment strategies and infection outcomes across a broader range of participants.

DETAILED DESCRIPTION:
This is a domain within the RATIONAL Platform Trial to test the effectiveness and safety of prophylactic antibiotics as an alternative Ig replacement in patients who have not yet commenced Ig replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be receiving IVIg replacement at standard dose for prevention of bacterial infections due to hypogammaglobulinaemia for at least 6 consecutive months.
2. Patient is not eligible for trial of Ig cessation in the opinion of the treating clinician and local investigator.

Exclusion Criteria:

1. Prior or planned allogeneic haematopoietic stem cell transplantation.
2. Major infection (Grade 3 or higher) in preceding 3 months, and or current active infection requiring systemic antimicrobial treatment.
3. Previous splenectomy.
4. Known history of bronchiectasis.
5. Previous participation in this domain.
6. Treating team deems enrolment in the domain is not in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS). | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Defined as time from randomisation (or, in domains with a single treatment arm, time from registration) until occurrence of a Grade 3 or higher infection (as defined by CTCAE Version 5), or death from any cause.

SECONDARY OUTCOMES:
Occurrence of at least one Grade 3 or higher infection(s) from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Occurrence of at least one Grade 3 or higher infection(s) from randomisation to 12 months.
Occurrence of one or more clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Occurrence of one or more clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months.
Number of clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Number of clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months.
Occurrence of one or more microbiologically documented infections from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Occurrence of one or more microbiologically documented infections from randomisation to 12 months.
Number of microbiologically documented infections from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Number of microbiologically documented infections from randomisation to 12 months.
All-cause mortality at 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  All-cause mortality at 12 months.
Infection-related mortality at 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Infection-related mortality at 12 months.
Time free from hospitalisation with antimicrobial administration with therapeutic intent from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Time free from hospitalisation with antimicrobial administration with therapeutic intent from randomisation to 12 months.
Occurrence of one or more treatment-related adverse events. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Occurrence of one or more treatment-related adverse events.
Number of treatment-related adverse events. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Number of treatment-related adverse events.
Isolation of fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Isolation of fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms from randomisation to 12 months.
Number of infections with fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms isolated from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Number of infections with fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms isolated from randomisation to 12 months.
Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months, using different questionnaire. | Randomisation, Month 3, Month 6, Month 9 and Month 12
  Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months, using different questionnaire.
Costs associated with allocated treatment arm and infections during study. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration).
  Costs of infections and trial interventions will be estimated based on trial treatment and adverse event data within the hospital medical record, as well as linked data obtained from the Medicare Benefits Scheme (MBS), Pharmaceutical Benefits Scheme (PBS) and Australian Immunisation Register (AIR). Data from the quality of life questionnaires will be used to calculate quality adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe McQuilten, Professor, Principal Investigator — Monash University
Locations (3):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Melbourne, Victoria
  - Northern Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available. Data will only be presented as a whole, no individual data will be published or presented.

REFERENCES:
- See also: Study Website — https://rationaltrial.com

DOCUMENTS (1):
  • Study Protocol (2023-11-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT07202065/Prot_000.pdf